CLINICAL TRIAL: NCT02538198
Title: Lenalidomide Maintenance in Plasma Cell Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-129
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Plasma Cell Myeloma
Keywords: lenalidomide (CC-5013); maintenance; 15-129
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

ARMS (1):
- Lenalidomide (Experimental): Subjects will receive lenalidomide 10 mg by mouth daily on days 1-21 of a 28-day cycle. Subjects may continue lenalidomide until disease progression, diagnosis of new malignancy, unacceptable toxicity, investigator discretion, voluntary withdrawal, or the end of the study (5 years); whatever comes first. Patients who complete at least four cycles of treatment will be considered evaluable.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide

SUMMARY:
This is a Phase 2 study to assess the good and bad effects of maintenance therapy on patients who have been treated for myeloma and no longer show signs of this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plasma cell myeloma treated with induction therapy or re-induction therapy, who at the time of study enrollment have documented evidence of stable disease response or better according to International Myeloma Workshop Consensus Panel
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of lenalidomide in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials
* ECOG performance status ≤ 2
* Patient must have adequate hematologic, renal, and hepatic, and as defined by:
* Absolute neutrophil count ≥ 1.0K /μL (growth factor support is permissible)
* Platelets ≥ 75K/μL (transfusions are permissible)
* Hemoglobin ≥ 8 g/dL (transfusions are permissible)
* Creatinine clearance (CrCl) of greater than or equal to 40 mL/min. using the CKD-EPI formula (see Appendix C). If the CrCl based on the CKD-EPI formula is <40 mL/min, the patient will have a 24 hr urine collection to measure CrCl. The measured CrCl must also be ≥ 40 ml/min.
* Total bilirubin ≤ 2 mg/dL, AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of childbearing potential* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS®) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.

  *A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).
* Females of childbearing potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy. See Appendix B: Lenalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Patients must be able to take daily prophylactic anticoagulation medication, such as: aspirin (81 or 325 mg) warfarin low molecular weight heparin or other medications as clinically indicated.
* Patient must understand and voluntarily sign an informed consent form, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Patients with progressive or refractory plasma cell myeloma, as defined by International Myeloma Workshop Consensus Panel criteria.
* Refractory to lenalidomide in the most recent line of therapy, as defined by the International Myeloma Consensus Panel criteria [47]- as failure to achieve minimal response or development of progressive disease while on lenalidomide or within 30 days of lenalidomide therapy
* Patients who are receiving any other investigational agents with the intent to treat myeloma. Permitted concurrent therapies include:
* Bisphosphonates
* Plasma cell leukemia
* Pregnant or breastfeeding females. Because there is a potential risk for adverse events to nursing infants secondary to treatment of the mother with lenalidomide, lactating females must agree not to breast feed while taking lenalidomide.
* Uncontrolled hypertension or diabetes
* Active hepatitis B or C infection
* Diagnosed or treated for another malignancy within 3 years prior to study enrollment, with the exception of complete resection of non-melanoma skin cancer, or an in situ malignancy.
* Previous diagnosis of another malignancy with any evidence of residual disease
* Patients seropositive for the human immunodeficiency virus (HIV), and/or those who are taking anti-retroviral treatment for HIV/AIDS.
* Prior organ transplant requiring immunosuppressive therapy
* Prior allogeneic stem cell transplant
* Patients requiring continuous, systemic immunosuppressive therapy
* Patients with myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled cardiac arrhythmias, or electrocardiographic evidence of acute ischemia
* Patients with conditions that would prevent absorption of the study drug
* Uncontrolled intercurrent illness including but not limited to uncontrolled infection or psychiatric illness/social situations that would compromise compliance with study requirements
* Significant neuropathy ≥Grade 3 at baseline
* Contraindication to concomitant anticoagulation prophylaxis
* Major surgery within 1 month prior to enrollment
* Patients who were previously exposed and who developed severe adverse events, hypersensitivity or desquamating rash to either thalidomide or lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years
  PFS is defined as time of start of treatment to time of progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lesokhin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Diamond B, Korde N, Lesokhin AM, Smith EL, Shah U, Mailankody S, Hultcrantz M, Hassoun H, Lu SX, Tan C, Rustad EH, Maura F, Maclachlan K, Peterson T, Derkach A, Devlin S, Landau HJ, Scordo M, Chung DJ, Shah GL, Lahoud O, Thoren K, Murata K, Ramanathan L, Arcila ME, Ho C, Roshal M, Dogan A, Giralt SA, Landgren O. Dynamics of minimal residual disease in patients with multiple myeloma on continuous lenalidomide maintenance: a single-arm, single-centre, phase 2 trial. Lancet Haematol. 2021 Jun;8(6):e422-e432. doi: 10.1016/S2352-3026(21)00130-7. PMID 34048681
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/